CLINICAL TRIAL: NCT04756245
Title: The Virtually Engaging Socially With Physical Activity (VESPA) Pilot Study
Brief Title: The VESPA Pilot Study
Acronym: VESPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Wells Fargo Faculty Scholar Endowment (Unknown)
Responsible Party: Principal Investigator, Jason Fanning, Assistant Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00023881
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Exercise; Behavior; Loneliness; Social Isolation
Keywords: Telehealth; Virtual Reality; Physical Activity
MeSH Terms: conditions — Motor Activity; Behavior; Social Isolation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two 4-week interventions: a virtual-reality or video conference-based group-mediated activity program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Participants engage in intervention procedures using virtual reality software.
  Interventions: Behavioral: Virtual Reality
- Video Conference (Active Comparator): Participants engage in intervention procedures using video conference software.
  Interventions: Behavioral: Video Conference

INTERVENTIONS:
Behavioral: Virtual Reality — Participants in this arm participate in 4 group-based behavioral counseling sessions plus 8 one-on-one coaching session within virtual reality software. Participants aim to engage in approximately 150 minutes per week of moderate-to-vigorous activity, with options including both virtual reality and real-world physical activities.
  Arms: Virtual Reality
Behavioral: Video Conference — Participants in this arm participate in 4 group-based behavioral counseling sessions plus 8 one-on-one coaching session within video conference software. Participants aim to engage in approximately 150 minutes per week of moderate-to-vigorous activity, with options including both streaming video and real-world physical activities.
  Arms: Video Conference

SUMMARY:
Physical activity has been described by the US federal government as a 'best buy' for public health. Unfortunately, most adults in the United States are not sufficiently active, and this worsens with age. Low levels of participation are driven by many challenging barriers, including lack of access, few opportunities for enjoyable activity, and few supportive social relationships, which is especially important given the central role of social connection for lasting behavior change.

A half-century of research in behavioral sciences has generated effective group-based physical activity programs, but these are inaccessible to most as they are often delivered in a few select research centers. Recent advances in telehealth have offered media for extending these interventions more broadly, but the experience of such programs is often hampered by technology that does not allow for a sense of physical and social presence. Fortunately, uptake of virtual reality (VR) is increasing rapidly, and the medium has a high level of potential for advancing the delivery of immersive evidence-based group interventions to those that most need it. Thus our specific aims are:

Specific aim 1: To test the feasibility and acceptability of a group-mediated physical activity intervention delivered fully via modern VR to older adults.

Specific aim 2: To examine the impact of this program on overall physical activity among older adults compared to the current standard-of-care for telehealth: the video conference meeting platform.

ELIGIBILITY:
Inclusion Criteria:

* Age of 45-80 years
* Body mass index between 30-45 kg/m2
* Low-active (30 or more minutes of moderate intensity physical activity on 2 or fewer days per week)
* Have access to home Wi-Fi
* Have regular access to a computer, tablet, or smartphone to receive teleconferencing calls
* Have a clear "VR space" (7'x7' object-free space)
* Have an "Activity buddy" (spouse, child, caregiver, etc.)
* Modified Telephone Interview for Cognitive Status (TICS-M) score of 32 or greater
* Consent from a physician for study participation
* Proficient in the English language
* Willingness to create or use existing personal Facebook account for virtual reality activities.

Exclusion Criteria:

* Current involvement in other physical activity research studies
* Hearing or sight impairments (significant visual or hearing impairment that cannot be corrected and results in the inability to use the telephone or hear normal conversation, colorblindness)
* Dependence on a cane or walker
* More than 1 fall in the past year
* Contraindication to exercise
* Current or recent history within the last 6 months of: symptomatic coronary heart disease, cancer, liver or renal disease, severe pulmonary disease, gross physical impairment, or uncontrolled hypertension; myocardial infarction or cardiovascular procedure within the last 3 months
* History of or diagnosis of photosensitive epilepsy
* Score of "severe" on any question in the Virtual Reality Sickness Questionnaire;
* Unwillingness to use a head-mounted virtual reality system
* Current severe or untreated depression

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of individuals attending all one-on-one and group calls | Weeks 0 through 4
  Feasibility will be assessed based on percentage of individuals attending all one-on-one and group calls
Acceptability | Baseline
  Percentage of individuals reporting no severe symptoms in response to virtual reality on the virtual reality sickness questionnaire

SECONDARY OUTCOMES:
Physical Activity | Baseline, Week 4
  Average daily steps over one week as recorded via Garmin VivoSmart 4
Social Relatedness | Baseline, Week 4
  Score on the social relatedness subscale of the Brief Psychological Needs Satisfaction and Frustration Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fanning, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kershner K, Morton D, Robison J, N'dah KW, Fanning J. Assessing the Feasibility and Acceptability of Virtual Reality for Remote Group-Mediated Physical Activity in Older Adults: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Nov 8;8:e53156. doi: 10.2196/53156. PMID 39514256